CLINICAL TRIAL: NCT06691451
Title: Inherited Thrombophilia and Thrombotic Risks in Inflammatory Bowel Disease During Activity and Remission
Brief Title: Inherited Thromophilia and Thrombotic Risks in Inflammatory Bowel Disease During Activity and Remission
Status: Not yet recruiting | Type: Observational
Sponsor: Asmaa mohammed abdelaal abdelaal (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Asmaa mohammed abdelaal abdelaal, Dr Asmaa Abdelaal, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Thrombophilia in ibd patients
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inherited thombopllia and thrombotic risks in inflammatory bowel Disease during activity and remission

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are systemic conditions characterized by multiple intestinal and extra-intestinal manifestations related to the associated chronic inflammatory state. Among their diverse extra-intestinal complications, venous thromboembolism (VTE) remains one of the most under recognized causes of morbidity and mortality in these patients, highlighting the need for a better understanding of the underlying mechanism of hypercoagulability, in addition to the role of acquired and inherited risk factors that further increase the risk of thrombosis with its impact on patients' outcomes.[1, 2]

ELIGIBILITY:
Inclusion Criteria:

* Age (18yrs - 65yrs) both sex

Exclusion Criteria:

* Presence of acquired cause (pregnancy, recent surgery, history of drug, History of malignant Disease, History of blood or blood product transfusion in last 4 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will be conducted at internal medicine department Assiut universty
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between the number of IBD patients with tendency to thrombosis in cases of activity- | Baseline
  -investigate the presence of multiple mutations associated with IBD patients with or without vascular complications.

REFERENCES:
- [Result] Yazici A, Senturk O, Aygun C, Celebi A, Caglayan C, Hulagu S. Thrombophilic Risk Factors in Patients With Inflammatory Bowel Disease. Gastroenterology Res. 2010 Jun;3(3):112-119. doi: 10.4021/gr2010.06.209w. Epub 2010 May 20. PMID 27942288